CLINICAL TRIAL: NCT01706393
Title: Double Blind Placebo Controled Randomized Trial, Effects of Probiotics Supplementation on Intestinal Microbiome in Malignancy Patients Who Get Pelvic/Abdominal Radiotherapy
Brief Title: Effects of Probiotics Supplementation on Intestinal Microbiome in Malignancy Pts(Get Pelvic/Abdominal Rtx)
Acronym: RTxIMprobio
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: SNUH-Cell-01
Record Dates: First submitted 2012-08-31; First posted 2012-10-15 (Estimated); Last update posted 2013-04-19 (Estimated); Status verified 2013-04

CONDITIONS: Cancer
Keywords: probiotics; intestinal microbiome; radiotherapy
MeSH Terms: conditions — Neoplasms | interventions — Probiotics

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- probiotics (Experimental): Probiotics supplementation group. Probiotics intake for 6 weeks(including 5weeks of Rtx) and it take one tablet twice a day.
  Probiotics is composed of Lactobacillus acidophilus, Streptococcus thermophilus, Bifidobacterium lactis, L. rhamnosus, B. longum and B. bifidum.
  Interventions: Dietary Supplement: probiotics (six probiotic cultures)
- placebo (Placebo Comparator): Placebo group. Placebo intake for 6 weeks(including 5weeks of Rtx) and it take one tablet twice a day.
  Placebo is composed of starch.Probiotics and placebo were similar in appearance, taste.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: probiotics (six probiotic cultures) — Effects of probiotics supplementation on intestinal microbiome; 2capsule bid orally for six weeks, 1capsule(500mg) Started eating probiotics one week prior of radiation therapy.
  Arms: probiotics
Dietary Supplement: Placebo — Placebo intake for 6 weeks(including 5weeks of Rtx) and it take one tablet twice a day.
  Arms: placebo

SUMMARY:
The purpose of this study is to evaluate the effect of probiotics to improve the intestinal microbiome in malignancy patients who get pelvic/abdominal radiotherapy.

DETAILED DESCRIPTION:
Pelvic/abdominal radiotherapy carries a risk of complications. Acute complications include diarrhea, abdominal pain, inflammatory change in the small intestine. Radiation creates changes in bacterial microbiome, the vascular permeability of the mucosal cells and in intestinal motility. Probiotics were known to improve gastrointestinal function. This is a randomized, double-blind, placebo-controlled study involving 26 patients designed to evaluate the effect of probiotics to change the intestinal microbiome in in patients undergoing concurrent pelvic/abdominal RT.

ELIGIBILITY:
Inclusion Criteria:

* Patients who current diagnosis of gynecologic cancer or rectal cancer and never previously received radiation therapy and will use for the first time radiotherapy at department of radiation oncology, Seoul National University Hospital.
* ECOG performance status (PS) of 0, 1, or 2.
* signed written informed consent.
* Patients who get pelvic/abdominal radiotherapy.

Exclusion Criteria:

* People who use antibiotics that can affect intestinal microorganism growth within one month before the study.
* Patients who use probiotics within one month before the study.
* Patients received neoadjuvant chemotherapy.
* Acute enteritis symptoms (diarrhea, abdominal pain, nausea, vomiting) for the patient.
* Patients diagnosed with inflammatory bowel disease.
* Patients suspected gastrointestinal infections and other infectious diseases.
* Suspected infections from blood tests : Excessive rise in WBC, ESR, CRP
* Suspected renal insufficiency from blood tests

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Estimated)
Dates: Start 2012-10; Primary Completion 2013-07 (Estimated); Study Completion 2013-07 (Estimated)

PRIMARY OUTCOMES:
Changes of gut microbial communities in malignancy patients receiving pelvic/abdominal radiotherapy after probiotics administration to prevent radiation enteropathy. | 42 days
  * Comparison of overall microbial communities in fecal samples between probiotics treated patients and control cancer patients receiving radiation therapy.
  * To determine preventing effect of probiotics against radiation enteropathy, all the bacterial species level taxon derived from fecal samples of cancer patients will be identified by massive sequencing analysis and relative abundance of each taxon between two groups will be statistically compared.
  * In addition, overall microbial composition, kind of species and their abundance, in two groups will be compared with clustering method such as UPGMA and PCoA and the variation values between two groups will be calculated.
  * In the current study, we will determine the effectiveness of probiotics for the prevention of radiation induced complications with these two comparative analysis methods.

SECONDARY OUTCOMES:
Prevention of any grade of diarrhea and gastrointestinal symptoms | 42 days
  * Gastrointestinal symptoms will be scored according the Gastrointestinal symptom rating scale before and after RTx.
  * Diarrhea will be graded weekly according the Common Toxicity Criteria system.

CONTACTS AND LOCATIONS:
Overall Officials: Hak Jae Kim, MD, Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea